CLINICAL TRIAL: NCT01044836
Title: A Randomized, Double-blind, Single-dosing, Crossover Study to Compare the Safety and Pharmacokinetic Characteristics of HD203 25 mg With Those of Enbrel® Injection 25 mg After Subcutaneous Injection in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetic Characteristics of HD203 in Healthy Male Volunteers
Acronym: SPH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanwha Chemical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EAGLE-I-09
Record Dates: First submitted 2010-01-05; First posted 2010-01-08 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Healthy volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental)
  Interventions: Biological: HD203

INTERVENTIONS:
Biological: HD203 — Injectable form

SUMMARY:
The purpose of this study is compare the safety and pharmacokinetic characteristics of HD203 with those of etanercept after subcutaneous injection in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years of healthy volunteers

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Etanercept levels in blood | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea